CLINICAL TRIAL: NCT05738304
Title: One-Day External Ureteral Catheter Versus Double-J Internal Ureteral Stent After Retrograde Intrarenal Surgery for Renal Stones: A Prospective, Randomized Trial
Brief Title: Ureteral Stenting After Retrograde Intrarenal Surgery for Renal Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abul-fotouh Ahmed, Professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uro_Azhar_11_023
Record Dates: First submitted 2023-02-11; First posted 2023-02-22 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Kidney Stone; Retrograde Intrarenal Surgery; Ureteral Stent
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Ureteral Catheter group (Experimental): After RIRS, an external ureteral catheter will be placed for one day.
  Interventions: Procedure: Retrograde intrarenal surgery with external ureteral catheter
- Double J group (Active Comparator): After RIRS, a double J internal ureteral stent will be placed for 2 weeks.
  Interventions: Procedure: Retrograde intrarenal surgery with double J internal ureteral stent

INTERVENTIONS:
Procedure: Retrograde intrarenal surgery with external ureteral catheter — The retrograde fURS sheathless technique will be used in all cases, including (a) cystourethroscopy with the introduction of a guidewire into the ipsilateral ureter up to the collecting system; (b) Semi-rigid ureteroscopy (using 9.5 Fr, Karl Storz, semi-rigid ureteroscope) for visualization of the ureter for any abnormalities, the introduction of the second guidewire and hydrophilic ureteral dilation; (c) introduction of the flexible ureteroscope (8.6 Fr, single-use digital flexible ureteroscope, OUT Medical Inc.) over the guidewire up to the kidney; (d) removal of the working guidewire after visualization of the stone; and (e) fragmentation of the stone using a holmium YAG laser device. All procedure steps will be performed under direct visualization and fluoroscopy guidance. At the end of the procedure, an external ureteral catheter will be placed for 24 hours.
  Arms: External Ureteral Catheter group
Procedure: Retrograde intrarenal surgery with double J internal ureteral stent — The retrograde fURS sheathless technique will be used in all cases, including (a) cystourethroscopy with the introduction of a guidewire into the ipsilateral ureter up to the collecting system; (b) Semi-rigid ureteroscopy (using 9.5 Fr, Karl Storz, semi-rigid ureteroscope) for visualization of the ureter for any abnormalities, the introduction of the second guidewire and hydrophilic ureteral dilation; (c) introduction of the flexible ureteroscope (8.6 Fr, single-use digital flexible ureteroscope, OUT Medical Inc.) over the guidewire up to the kidney; (d) removal of the working guidewire after visualization of the stone; and (e) fragmentation of the stone using a holmium YAG laser device. All procedure steps will be performed under direct visualization and fluoroscopy guidance. At the end of the procedure, a double-J internal ureteric stent will be placed for 2 weeks.
  Arms: Double J group

SUMMARY:
Several studies evaluated the benefit of a short-term external ureteral catheter (UC) compared to double-J (DJ) ureteral stent after flexible ureteroscopy (URS); the results were controversial. These studies had combined analyses of ureteral and renal stones with a high risk of selection bias. Studies comparing external UC and DJ stent after flexible URS for isolated renal stones are lacking.

In the present study, the investigators will compare the outcomes of using a one-day external UC versus a DJ internal ureteral stent for ureteral drainage after retrograde flexible URS (retrograde intrarenal surgery "RIRS") for renal stones. The investigators aim to identify the best ureteral drainage method after RIRS regarding stone clearance, complications, and stent-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients of either gender in whom RIRS was the primary modality.

Exclusion Criteria:

* Pregnant women
* Active urinary tract infection
* solitary kidney
* Concomitant pathology that need intervention in the same setting
* Patients with surgical incidents that indicate double-J stenting (Residual sizable fragments, ureteral false passage, ureteral mucosal laceration, ureteral perforation, and calyceal rupture).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | up to 1 month
  No stones or residual fragments >3 mm on postoperative imaging study
Stent-related symptoms | from post operative day one till double J removal; an average of 2 weeks
  Irritative lower urinary tract symptoms

SECONDARY OUTCOMES:
Postoperative renal pain | up to 1 month
  Renal pain attacks and severity as evaluated by visual analogue pain scale (VAPS).
  The VAPS is a pain rating scale based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
Rehospitalization rate | From post RIRS home discharge up to one month
  the need for unscheduled hospital admission
Reintervention rate | up to 3 months
  the need for reoperation

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Department, Al-Azhar University Hospital, Cairo, Egypt